CLINICAL TRIAL: NCT03704311
Title: Evaluation of Mitochondrial Function in Chronic Myofascial Trigger Points - A Prospective Cohort Pilot Study Using High-resolution Respirometry
Brief Title: Evaluation of Mitochondrial Function in Myofascial Trigger Points Cohort Pilot Study Using High-resolution Respirometry
Acronym: MitoTrigger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MUInnsbruck
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Pain, Neck; Pain, Back; Myofascial Trigger Point Pain; Myofascial Pain; Mitochondrial Pathology
MeSH Terms: conditions — Neck Pain; Back Pain; Myofascial Pain Syndromes

STUDY DESIGN:
Masking Description: Assessor doing high Resolution respirometry was blinded with respect to diagnosis, location of biopsy and all Patient related data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Experimental): Evaluation of mitochondrial function after muscle biopsy and follow-up for surgical complications.
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy — Local anesthesia was applied to the superficial skin covering the MTrP of each participant. Percutaneous biopsy sampling optimized with a suction-enhancement technique was used to obtain muscle biopsies of the m. trapezius MTrP or the m. gluteus medius MTrP from each participant using small Bergstrom muscle biopsy needle, 8 swg (4.0mm) x 100 mm (Dixons Surgical Instruments, Essex, United Kingdom).

SUMMARY:
This pilot study established a minimally invasive biopsy technique to obtain high-quality MTrP tissue samples to evaluate mitochondrial function via high-resolution respirometry.

DETAILED DESCRIPTION:
Myofascial trigger points (MTrPs) are hyperirritable areas in the fascia of the affected muscle, possibly related to mitochondrial impairment. They can result in pain and hypoxic areas within the muscle. This pilot study established a minimally invasive biopsy technique to obtain high-quality MTrP tissue samples to evaluate mitochondrial function via high-resolution respirometry. Secondary objectives included the safety of the biopsy procedure assessed via clinical wound healing (number of patients with signs for local infection and inflammation). For this purpose, twenty healthy males participated in this study, 10 with a diagnosis of myofascial pain in the musculus (m.) trapezius MTrP (TTP group) and 10 with a diagnosis of myofascial pain in the m. gluteus medius (GTP group). The affected muscle was biopsied followed by a biopsy from the vastus lateralis to be used as a control. Measurements of oxygen consumption were carried out using high-resolution respirometry.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18-45 years
* Clinical diagnosis of myofascial pain syndrome within the region of the shoulder-neck muscles or the lumbogluteal region and the presence of an MTrP, defined as a firm palpation of a hard, tender nodule resulting in a spontaneous pain complaint
* with symptoms present for 1 to 12 months

Exclusion Criteria:

* Signs that the participant's prescriptive compliance was not expected (e.g., lack of cooperation)
* Disorders of the respiratory tract
* Neurological disorders, in particular neurodegenerative and neuromuscular diseases
* Disorders of the cardiovascular system or the musculoskeletal system
* Civil servants and military service personnel.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Mitochondrial function in myofascial trigger points | Baseline measurement
  Mitochondrial respiration was assessed from muscle biopsy samples obtained from trigger points of the musculus trapezius and the musculus gluteus medius

SECONDARY OUTCOMES:
Number of participants with biopsy-related impaired wound healing | Baseline and follow-up assessment (1 week after the baseline biopsy)
  Clinical wound assessment (number of patients with signs for local infection and inflammation)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Fischer, MD, PhD, Principal Investigator — Medical University Innsbruck

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fischer MJ, Horvath G, Krismer M, Gnaiger E, Goebel G, Pesta DH. Evaluation of mitochondrial function in chronic myofascial trigger points - a prospective cohort pilot study using high-resolution respirometry. BMC Musculoskelet Disord. 2018 Oct 30;19(1):388. doi: 10.1186/s12891-018-2307-0. PMID 30376863